CLINICAL TRIAL: NCT05880290
Title: Performance of the Gynaecological Examination in the Lateral Decubitus Position
Acronym: EXADELA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/0375/HP
Record Dates: First submitted 2023-03-21; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Medical Care

STUDY DESIGN:
Intervention Model Description: Single group: gynaecological examination in lateral decubitus, conventional repositioning if unsuccessful
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gynaecological examination in lateral decubitus, conventional repositioning if unsuccessful (Experimental)
  Interventions: Procedure: gynaecological examination in lateral decubitus

INTERVENTIONS:
Procedure: gynaecological examination in lateral decubitus — Single group: gynaecological examination in lateral decubitus, conventional repositioning if unsuccessful

SUMMARY:
The gynaecological examination consists of a breast examination, abdominal examination, inspection of the vulva, vaginal touch and pelvic examination with a speculum.

The latter is essential for the insertion and removal of intrauterine devices (IUDs), for the diagnosis and screening of pathologies that may cause pelvic symptoms, for assessment of the vaginal wall and for regular screening for cervical cancer.

The gynaecological examination is feared by many women because of the feeling of exposure, vulnerability and loss of control.

The parallel with a sexual position is particularly disturbing for patients who do not want to see this representation mixed with a medical necessity, which can lead some women to have irregular or even discontinued follow-up.

For the past ten years, medical practice theses and midwifery dissertations have evaluated the interest of another position for the pelvic examination with the speculum : the lateral decubitus position in which the patient lies on her side.

The lateral decubitus pelvic examination seems to be an alternative for comfort and respect for modesty, which is favoured by the patients.

This examination position would have advantages in situations of anterior anatomical position of the position of the cervix, prolapse, severe obesity, hip pathology or significant reluctance to the examination.

The effectiveness of this technique in terms of examination performance needs to be evaluated to promote its dissemination.

The impact of an examination that is better experienced by patients is that of better adherence and therefore better follow-up, which is the particular challenge of primary care.

Single group: gynaecological examination in lateral decubitus, conventional repositioning if unsuccessful

ELIGIBILITY:
Inclusion Criteria:

* Woman of legal age, 18 years or older.
* Who already had a gynaecological examination in the conventional position.
* Requiring a gynaecological consultation in primary care with speculum for screening, diagnosis or prevention.
* Woman of childbearing age with a negative urine pregnancy test or postmenopausal woman (no period in the last 12 months).
* Patient who has read and understood the information letter and signed the consent form.
* Affiliated to the social security.

Exclusion Criteria:

* Pregnant woman
* Who already participated to this protocol
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection / sub-guardianship or curatorship.
* Major cognitive impairment that prevents the subject from fully understanding the requirements for participation in the study or from giving informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Gynaecological speculum examination in the lateral decubitus position will be perform during the visit to assess if the performance is sufficient to be offered as an alternative to the examination in the conventional position. | 1 day
  Examination realize during the visit of the patient.

SECONDARY OUTCOMES:
Clinicians' satisfaction with lateral decubitus positioning for pelvic speculum examination will be evaluate with a questionnaire | 1 day
  The questionnaire will be completed by the investigator during each visit.
patients' satisfaction with lateral decubitus positioning for pelvic speculum examination will be evaluate with a questionnaire | 1 day
  The questionnaire will be completed by the patient during each visit.
The performance (success rate) of early examination (6 first examinations) will be evaluated for each practicioner. | 1 day
  Success rate in the first 6 patients of each practicioner. This result will allow us to know if the technique is accessible.
The occurrence of complications at 3 months during IUD insertion in the lateral position will be quantified | 3 months
  We will call each patient for follow-up at 3 months for patients with IUD insertion in the lateral position.
The predictive factors for failure of the lateral decubitus examination will be determined | 1 day
  Age (years), weight (kg) and reason for speculum exam (IUD placement, pelvic pain, vaginal discomfort) will be collected and correlated. This information will make it possible to define a population at risk of failure of the examination in lateral decubitus.